CLINICAL TRIAL: NCT00821067
Title: The Effect of Oral D-Ribose in "Baby Boomers" With Fatigue. A Randomized, Double-Blind Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioenergy Life Science, Inc. (Industry)
Responsible Party: Jeff Thompson, Bioenergy Life Science, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FS20081121
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Ribose; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): A 6 gm/day (3 gm/bid) dose of D-ribose
  Interventions: Dietary Supplement: D-ribose
- 2 (Placebo Comparator): A 6 gm/day (3 gm/bid) dose of dextrose.
  Interventions: Dietary Supplement: Dextrose

INTERVENTIONS:
Dietary Supplement: D-ribose — A 6 gm/day (3 gm/bid) dose of D-ribose in water. Each subject will consume oral D-ribose, dissolved in 8 fl. oz of water (1 serving) twice daily, for 2 weeks.
  Arms: 1
Dietary Supplement: Dextrose — A 6 gm/day (3 gm/bid) dose of dextrose in water. Each subject will consume oral dextrose, dissolved in 8 fl. oz of water (1 serving) twice daily, for 2 weeks.
  Arms: 2

SUMMARY:
D-ribose, a natural occurring pentose carbohydrate, has repeatedly shown to enhance high-energy phosphates and improve function following ischemia, states of congestive heart failure, and recently in subjects with lung disease. An initial preliminary, open label pilot study demonstrated a positive benefit of D-ribose in "Baby-Boomer" subjects aged 50 to 65 years old complaining of persistent fatigue. The objective of this study will build on the previously collected data to evaluate oral D-ribose vs. dextrose (administered as a supplement) in relatively healthy, yet fatigued subjects with a goal of improving their state of fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Presents with complaint of fatigue with duration longer than one month
* Males/Females between the ages of 50 and 65 years of age
* No previous clinical diagnosis of pulmonary, cardiac or metabolic disorders based on history
* Capable of performing a sub-maximal incremental treadmill exercise using cardiopulmonary analysis methods
* Normal blood pressure or those with mild, untreated pre-hypertension (>120/70 or < 140/90 mmHg)
* Able to be compliant with the supplement regimen, repeat clinical visits and completion of the study questionnaires
* Must be able to understand the consent form, agree to participate, and to execute their signature

Exclusion Criteria:

* Not presently taking any adenine nucleotide enhancing supplements
* History of non-compliance in previous studies
* Known to be pregnant
* Uncontrolled cardiac arrhythmias causing symptoms or unstable hemodynamics
* Moderate to severe gout
* A diagnosis of arthritis of the lower extremities
* Mental impairment, inability to cooperate
* History of acute non-cardiopulmonary disorder that may affect exercise performance, (e.g. infection, renal failure, thyrotoxicosis, etc.)
* Any disorder or condition that in the opinion of the study physician would render exercise unsafe or would impact exercise performance
* Any person who is incarcerated, or on a work release program

Additional Exclusions observed and sequelae during initial baseline evaluation:

* Drop in systolic blood pressure of >10 mm Hg from baseline despite an increase in workload, when accompanied by other evidence of ischemia
* Moderately severe angina
* Increasing nervous system symptoms (e.g. ataxia, dizziness, or near syncope)
* Signs of poor perfusion (cyanosis or pallor)
* Technical difficulties monitoring the ECG or systolic blood pressure
* Subject's desire to stop
* Sustained ventricular tachycardia
* Electrocardiographic ST elevation (+1.0 mm) in leads without diagnostic Q-waves (other than V1 or aVR)

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
CPX parameters relative to placebo as measured by: | Two weeks
VO2 at AT | Two weeks
Ventilation Efficiency Slope | Two weeks
Oxygen Uptake Efficiency Slope | Two weeks
Heart rate to METS ratio at AT | Two weeks
Net Energy Expenditure at AT | Two weeks

SECONDARY OUTCOMES:
The secondary objective will be to subjectively evaluate the subjects' level of fatigue and will be assessed by a serial questionnaire. | Two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Aurora Denver Cardiology Association, Denver, Colorado, United States